CLINICAL TRIAL: NCT02924961
Title: Fluoroscopic and RSA Evaluation of the Triathlon Total Knee Prosthetic Design
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Mobile-bearing insert dislocation
Sponsor: Leiden University Medical Center (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Principal Investigator, R.G.H.H. Nelissen, Prof. dr., Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P07.205
Record Dates: First submitted 2016-09-21; First posted 2016-10-05 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Complications; Arthroplasty, Mechanical; Aseptic Loosening

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triathlon Mobile-bearing (Experimental): Primary total knee replacement with cemented Triathlon posterior stabilized mobile-bearing
  Interventions: Device: Triathlon PS total knee system with mobile-bearing
- Triathlon Fixed-bearing (Active Comparator): Primary total knee replacement with cemented Triathlon posterior stabilized fixed-bearing
  Interventions: Device: Triathlon PS total knee system with fixed-bearing

INTERVENTIONS:
Device: Triathlon PS total knee system with mobile-bearing
  Other Names: Stryker Orthopaedics
  Arms: Triathlon Mobile-bearing
Device: Triathlon PS total knee system with fixed-bearing
  Other Names: Stryker Orthopaedics
  Arms: Triathlon Fixed-bearing

SUMMARY:
The goal of this study is to compare the fixed bearing (FB) Triathlon knee (Stryker, USA) and the mobile bearing (MB) Triathlon knee (Stryker, USA) and study the effect of implant design on kinematics and micromotion. During two tasks the kinematics measured with fluoroscopy (kinematics and movement of the polyethylene bearing). Roentgen Stereophotogrammetric Analysis (RSA) will be used to evaluate micromotion between prosthesis and the bone for the MB and FB Triathlon knee.

DETAILED DESCRIPTION:
The goal of this study is to perform a kinematic evaluation of a MB and FB knee prosthesis designs (Triathlon, Stryker, USA), by means of fluoroscopy and RSA and compare the different designs. The findings of this study will contribute to improve total knee designs and improve rehabilitation strategies.

Objectives:

1. To evaluate if there is micromotion of the prosthesis with respect to the bone and if there is a different migration pattern between the designs.
2. To assess and compare the in vivo kinematic patterns of the knee designs by means of fluoroscopy. This will be done on a subset of the patients (the first 20 patients able to perform step-up and lunge motions 6 months post-operatively in a controlled manner without the use of bars and walk more than 1 km)
3. To evaluate if the polyethylene bearing in the mobile bearing is rotating and if this changes over time.
4. Results of the RSA study will be used to correlate the kinematic parameters (fluoroscopy) with the migration results in order to identify factors of risk for the survival of total knee prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Patient (minimum age of 18 years old, no maximum age limit) is diagnosed with osteoarthritis or rheumatoid arthritis and requires primary arthroplasty.
* Patient is capable of giving informed consent and expressing a willingness to comply with this study
* Patient has no major deformities (i.e. sagittal and coronal deformities are less then 15 degrees)
* The ability to perform a lunge and step-up motion without the help of bars or a cane.
* No or slight pain during activity according to the Knee Society Pain Score

Exclusion Criteria:

* The patient is unable or unwilling to sign the Informed Consent specific to this study
* The individual has a functional impairment of any other lower extremity joint besides the operated knee
* Patient has a flexion contracture of 15° and more
* Patient has a varus/valgus contracture of 15° and more
* Patients requiring revision arthroplasty
* The patient does not understand the Dutch or English language good enough to participate.
* The use of walking aids
* The inability to walk more than 500 meters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-04; Primary Completion 2011-07 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Migration, measured by means of RSA on the first 20 patients (fluoroscopy subset) | First or second day postoperatively, 6 months, 1 year
  Migration (MTPM in mm) of the prosthesis with respect to the host bone measured by means of roentgen stereophotogrammetric analysis (RSA)

SECONDARY OUTCOMES:
Migration, measured by means of RSA | First or second day postoperatively, 6 months, 1 year and annually thereafter up to 20 years
  Migration (MTPM in mm) of the prosthesis with respect to the host bone measured by means of roentgen stereophotogrammetric analysis (RSA)
Assessment of the knee flexion range by means of fluoroscopy during step-up motions | 6 months and 13 months postoperatively
  Patients will be asked to perform three step-up motions (height 18 cm) with bare feet in front of a flat panel fluoroscope. Outcome measurement is knee flexion range (degrees).
Assessment of the axial rotation range of femoral component by means of fluoroscopy during step-up motions | 6 months and 13 months postoperatively
  Patients will be asked to perform three step-up motions (height 18 cm) with bare feet in front of a flat panel fluoroscope. Outcome measurement is axial rotation range of femoral component (degrees).
Assessment of the knee flexion range by means of fluoroscopy during lunge motions | 6 months and 13 months postoperatively
  Patients will be asked to perform three lunge motions (height 18 cm) with bare feet in front of a flat panel fluoroscope. Outcome measurement is knee flexion range (degrees).
Assessment of the axial rotation range of femoral component by means of fluoroscopy during lunge motions | 6 months and 13 months postoperatively
  Patients will be asked to perform three lunge motions (height 18 cm) with bare feet in front of a flat panel fluoroscope. Outcome measurement is axial rotation range of femoral component (degrees).
Investigation of clinical performance and patient outcome with the Knee Society Score (KSS) | Within 3 months prior to surgery, 6 months postoperatively, 1 year and and annually thereafter up to 20 years
  The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, range of motion (ROM) and joint stability, and one for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: R.G.H.H. Nelissen, MD, PhD, Principal Investigator — Head of Department of Orthopaedics, Leiden University Medical Center
Locations (1):
- Department of Orthopaedics, Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
IPD analysis is scheduled